CLINICAL TRIAL: NCT01871558
Title: Randomized, Open-label, SU-controlled Study of 24-week Duration to Compare Metformin/Vildagliptin + Basal Insulin Versus Metformin/SU + Basal Insulin in T2DM Patients Starting Basal Insulin After Failing Metformin/SU
Brief Title: Vildagliptin/Metformin in T2DM Patients Starting Basal Insulin
Acronym: ADDONIS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CLAF237AFR07
Record Dates: First submitted 2013-06-04; First posted 2013-06-06 (Estimated); Results first posted 2016-03-23 (Estimated); Last update posted 2016-04-21 (Estimated); Status verified 2016-03

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: type 2 diabetes; basal insulin; vildagliptin
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Vildagliptin; Metformin; Sulfonylurea Compounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- SU+metformin + Basal Insulin (Active Comparator): Randomized patient will remain on their previous dual therapy by SU+metformin, which will be kept unchanged, + start of Basal Insulin up-titrated as per usual algorithms primarily based on FPG
  Interventions: Drug: Metformin; Drug: sulfonylurea (SU); Drug: Basal Insulin
- Metformin/vildagliptin + Basal Insulin (Experimental): Randomized patient will receive Vildagliptin 50 mg twice daily (b.i.d) + continued therapy with Metformin, + start of Basal Insulin up-titrated as per usual algorithms primarily based on FPG
  Interventions: Drug: Vildagliptin; Drug: Metformin; Drug: Basal Insulin

INTERVENTIONS:
Drug: Vildagliptin — 50 mg b.i.d
  Other Names: Galvus
  Arms: Metformin/vildagliptin + Basal Insulin
Drug: Metformin — metformin is to be kept unchanged
Drug: sulfonylurea (SU)
  Arms: SU+metformin + Basal Insulin
Drug: Basal Insulin

SUMMARY:
To compare a therapeutic strategy combining vildagliptin+metformin + Basal Insulin versus SU+metformin + Basal Insulin on the incidence of hypoglycemic events over 24 weeks.

DETAILED DESCRIPTION:
This study, conducted in T2DM patients failing a dual therapy with metformin/SU in whom the decision to start basal insulin has been taken, will compare vildagliptin+metformin versus the previously used SU+met combination (regimen kept unchanged) in association with basal insulin, up-titrated as per usual algorithms primarily based on FPG to obtain a similar improvement in glycemic control in both arms, on the incidence of hypoglycemic episodes over 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* T2DM patients inadequately controlled with metformin+ SU combination therapy at max tolerated doses and in whom the decision to start basal insulin has been taken
* with stable metformin+ SU combination therapy for at least 12 weeks prior to randomization
* with a glycemic target of HbA1c <= 7%
* with HbA1c at inclusion >7% and <=9%
* Patients willing and able to start basal insulin and perform appropriate self monitoring of blood glucose (SMBG)

Exclusion Criteria:

* contraindication for either SUs, metformin or insulin and history of hypersensitivity to vildagliptin
* acute or chronic diseases that interfere with efficacy/safety results of this trial or put patient at risk

Other protocol defined inclusion/exclusion criteria may apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-06; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (19):
- France (19):
  - Novartis Investigative Site, Antibes
  - Novartis Investigative Site, Auxerre
  - Novartis Investigative Site, Bar-le-Duc
  - Novartis Investigative Site, Bondy
  - Novartis Investigative Site, Brest
  - Novartis Investigative Site, Caen
  - Novartis Investigative Site, Corbeil-Essonnes
  - Novartis Investigative Site, Fleury-sur-Orne
  - Novartis Investigative Site, Maisons-Laffitte
  - Novartis Investigative Site, Menton
  - Novartis Investigative Site, Montpellier
  - Novartis Investigative Site, Paris
  - Novartis Investigative Site, Rennes
  - Novartis Investigative Site, Saint-Nazaire
  - Novartis Investigative Site, Sanary-sur-Mer
  - Novartis Investigative Site, Strsbourg
  - Novartis Investigative Site, Toulouse
  - Novartis Investigative Site, Valence
  - Novartis Investigative Site, Valenciennes

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Metformin/Vildagliptin + Basal Insulin | SU+Metformin + Basal Insulin
Started | 21 | 21
Completed | 18 | 19
Not Completed | 3 | 2
Not completed — Other reason | 0 | 1
Not completed — antidiabetic drug prematurely stopped | 1 | 1
Not completed — Withdrawal by Subject | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Metformin/Vildagliptin + Basal Insulin | SU+Metformin + Basal Insulin | Total
Number analyzed (Participants) | 21 | 21 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.6 (12.52) | 66.8 (7.80) | 63.7 (10.77)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 8 | 18
  Male | 11 | 13 | 24

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Who Reported at Least One Symptomatic Hypoglycemic Event During the 24 Week Randomized Period in Both Treatment Arms
Time Frame: 24 weeks
Population: safety population
Measure: Number; unit: percent of participants
Arm/Group | Metformin/Vildagliptin + Basal Insulin | SU+Metformin + Basal Insulin
Number analyzed (Participants) | 21 | 21
percent of participants | 22.2 | 45.0
Statistical Analysis 1: Comparison: Metformin/Vildagliptin + Basal Insulin vs SU+Metformin + Basal Insulin; Test type: Superiority or Other; p = 0.139, Chi-squared

2. Secondary Outcome: Percentage of Patients Reaching Their Glycemic Target Without Hypoglycemic Events
Description: Glycemic target is defined as Glycated hemoglobin(HbA1c) ≤ 7%
Time Frame: 24 weeks
Population: ITT population
Measure: Number; unit: percent of participants
Arm/Group | Metformin/Vildagliptin + Basal Insulin | SU+Metformin + Basal Insulin
Number analyzed (Participants) | 19 | 19
percent of participants | 44.4 | 47.4

3. Secondary Outcome: Change From Baseline in HbA1c to Week 24 in Both Treatment Arms
Time Frame: Baseline, Week 24
Population: ITT population
Measure: Mean (Standard Deviation); unit: HbA1c percent
Arm/Group | Metformin/Vildagliptin + Basal Insulin | SU+Metformin + Basal Insulin
Number analyzed (Participants) | 19 | 19
HbA1c percent
  baseline | 8.2 (0.56) | 8.2 (0.42)
  week 24 | 7.2 (0.71) | 7.4 (0.89)

4. Secondary Outcome: Change From Baseline in Body Weight in Both Treatment Arms
Time Frame: Baseline, Week 24
Population: Safety Population
Measure: Mean (Standard Deviation); unit: kg
Arm/Group | Metformin/Vildagliptin + Basal Insulin | SU+Metformin + Basal Insulin
Number analyzed (Participants) | 21 | 21
kg | -0.3 (2.51) | 1.4 (2.61)

5. Secondary Outcome: Mean Daily Insulin Dose at Week 24
Time Frame: Week 24
Population: ITT population
Measure: Mean (Standard Deviation); unit: (U/d)
Arm/Group | Metformin/Vildagliptin + Basal Insulin | SU+Metformin + Basal Insulin
Number analyzed (Participants) | 19 | 19
(U/d) | 33.0 (23.08) | 19.8 (13.83)

6. Secondary Outcome: Percentage of Patients With Severe and Confirmed Hypoglycemic Events
Description: Severe hypoglycemic events (and number of events) , defined as events requiring assistance of a third party, and with confirmed hypoglycemic events (and number of events) defined as events with concomitant self monitoring of blood glucose (SMBG) < 70 mg/dL
Time Frame: 24 weeks
Population: ITT population
Measure: Number; unit: percent participants
Arm/Group | Metformin/Vildagliptin + Basal Insulin | SU+Metformin + Basal Insulin
Number analyzed (Participants) | 19 | 19
percent participants | 0.0 | 0.0

7. Secondary Outcome: Percent of Participants That Reach Therapeutic Goal (HbA1c ≤ 7%) at Week 24 Without Any Hypoglycaemic Episode (Symptomatic or Not) and Without Any Weight Gain (Variation ≥3% Compared to Baseline)
Description: HbA1c <= 7% without any hypoglycaemic episode (symptomatic or not) and without any weight gain
Time Frame: week 24
Population: ITT population
Measure: Number; unit: percent of participants
Arm/Group | Metformin/Vildagliptin + Basal Insulin | SU+Metformin + Basal Insulin
Number analyzed (Participants) | 19 | 19
percent of participants | 27.8 | 21.1

ADVERSE EVENTS:
Arm/Group | Metformin/Vildagliptin + Basal Insulin | SU+Metformin + Basal Insulin
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/21
Other Adverse Events (participants affected / at risk) | 4/21 | 10/21
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Metformin/Vildagliptin + Basal Insulin (N=21) | SU+Metformin + Basal Insulin (N=21)
Conjunctival haemorrhage (Eye disorders) | 0 | 1
Visual impairment (Eye disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 2
Fatigue (General disorders) | 0 | 1
Injection site pain (General disorders) | 0 | 1
Tooth abscess (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 1
Wound (Injury, poisoning and procedural complications) | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Headache (Nervous system disorders) | 0 | 1
Parkinson's disease (Nervous system disorders) | 0 | 1
Sciatica (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Renal colic (Renal and urinary disorders) | 1 | 0
Cataract operation (Surgical and medical procedures) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.